CLINICAL TRIAL: NCT06389994
Title: Monitoring Eosinophilic Esophagitis During Food Oral Immunotherapy Using Esophageal String Test
Brief Title: Esophageal String Test Monitoring to Monitor Eosinophilic Esophagitis During Oral Immunotherapy
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Jonathan Spergel, Professor of Pediatrics; Chief, Allergy Section Director of Center for Pediatric Eosinophilic Disease, Children's Hospital of Philadelphia
Other Study IDs: 23-021041
Record Dates: First submitted 2024-04-19; First posted 2024-04-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing oral immunotherapy: All patients will have esophageal string test
  Interventions: Device: Esophageal String Test

INTERVENTIONS:
Device: Esophageal String Test — The EnteroTracker® capsule is supplied in pouches, each pouch containing a single capsule. The device is comprised of an ingestible capsule that contains a weighted ball and a highly absorbent nylon string. The looped portion of the string is secured externally to the patient's cheek and the rest of the capsule is swallowed by the patient.
  Other Names: EnteroTracker®

SUMMARY:
Patients with IgE mediated food Allergy have elevated risk of eosinophilic esophagitis, and new therapies like oral immunotherapy (OIT) carry additional risk of Eosinophilic Esophagitis (EoE). The goal of this study is to investigate the Esophageal String Test (EST) as a screening tool for Eosinophilic Esophagitis (EoE) during OIT therapy. Investigators will compare the efficacy of the Esophageal String Test to symptom assessment using a validated patient reported symptom questionnaire, the Pediatric Eosinophilic Esophagitis Symptom Score (PEESS) v2.0. Investigators will utilize these tools to screen patients at their baseline visit prior to the start of OIT, then at the 3- and 6-month OIT follow-up visits.

DETAILED DESCRIPTION:
The goal of this study is to investigate the EST as a screening tool for EoE during OIT therapy. Investigators will utilize these tools to screen patients at their baseline visit prior to the start of OIT, then at the 3- and 6-month OIT follow-up visits.

The primary objectives are to assess feasibility of the EST as a screening tool for EoE in IgE mediated food allergy patients in an OIT program.

The secondary objective(s) are to: (1) estimate the correlation of EST and PEESS in screening for EoE in IgE mediated food allergy patients in an OIT program, (2) provide an estimate of the prevalence of EoE in IgE mediated food allergy patients, which Investigators will measure at the time of presentation for OIT, (3) provide an estimate of the incidence of development of EoE during the first 3- and 6- months of OIT.

The study will take place at the Children's Hospital of Philadelphia Food Allergy Clinic sites that participate in OIT. There will be 75 participants ages 7-18 years of age with IgE mediated food allergy who are undergoing oral immunotherapy for food allergies.

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all of the following criteria:

* Male or female, aged 7 to 18 years old, inclusive
* Have a history of Immunoglobulin (IgE)-mediated food allergy
* Considering using oral immunotherapy (OIT) for food allergies at CHOP°
* Able & willing to swallow the esophageal capsule
* Parental/guardian permission (informed consent) and if appropriate, child assent.
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Known or expected need for MRI imaging during the study period
* Known connective tissue disease
* Known eosinophilic disorder including any eosinophilic gastrointestinal disorder and hypereosinophilic disorder
* Past history of caustic ingestion or other esophageal injury
* History of esophageal surgery or dilation (i.e.: tracheoesophageal fistula repair)
* History of gastrointestinal motility disorder including esophageal achalasia
* History of inflammatory bowel disease
* Unwilling or unable to swallow the EST
* Oral or intravenous steroids in the preceding 60 days (not including swallowed topical fluticasone, budesonide, etc.)
* Participation in a clinical study that may interfere with participation in this study
* Pregnant or lactating females
* Limited English proficiency
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 7 years of age or older with IgE mediated food allergy undergoing OIT at Children's Hospital of Philadelphia (CHOP) will be enrolled in this study. Prior work at CHOP and other pediatric centers has demonstrated that most children 7 years and older can swallow EST capsules.
  Subjects will be identified by reviewing the Electronic Medical Record of IgE-mediated food allergy patients scheduled for evaluation in CHOP Allergy Clinic OIT clinic. Informed consent and assent will be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-02 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Esophageal String Test | baseline, 3 month and 6 months
  Esophageal String Test (EST) will measure presence of eosinophilic protein. Higher score is more eosinophils.. Range is 0 to 100

SECONDARY OUTCOMES:
Prevalence of Eosinophilic Esophagitis | Baseline, 3 month and 6 months
  EOE will be determined by the upper endoscopy showing greater than 15 eos/hpf. Normal is zero. Range is from 0 to 100
Eosinophilic Esophagitis Symptoms | Baseline, 3 month and 6 months
  EOE symptoms will be measured by Pediatric Eosinophilic Esophagitis Symptom Score.
  HIgher score indicates more symptoms. Range is zero to 72

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Spergel, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) available to other researchers.